CLINICAL TRIAL: NCT03951701
Title: Evaluation of Interest of a Systematic Screening for Oncological Supportive Care
Brief Title: Evaluation of Interest of a Systematic Screening for Oncological Supportive Care Needs
Acronym: DBSOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-02; 2018-A01425-50 (Other: ANSM)
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Supportive Care Needs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- observation cohort (Experimental): Questionnaire to assess the supportive care needs
  Interventions: Other: Evaluation of the supportive care

INTERVENTIONS:
Other: Evaluation of the supportive care — Evaluation of interest of a systematic screening for oncological supportive care needs

SUMMARY:
Monocentric, descriptive, cross-sectional, interventional, prospective and non-randomized study.

DETAILED DESCRIPTION:
The study will unfold in the followed day hospital's departments of the Paul Strauss Cancer Center (Strasbourg, France) : supportive care department, chemiotherapy department and radiotherapy department. The study is based on two questionnaires that include six sections : nutrition, social, psychologic, physiotherapy, pain and supportive care needs evaluation.

The first questionnaire gives information about the patient and allow to screen supportive care needs. It should be read by medical or paramedical staff who report the function of the reader and options that are proposed to the patient after reading the questionnaire.

The second questionnaire will be done after 4 to 6 weeks by a phone call from the clinical research nurse. The objective of this questionnaire is to determine what kind of care have been provided.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for a cancer
* Age ≥ 18 years old
* Receiving treatment (chemotherapy and/or radiotherapy) in day hospital and/or supportive care department
* Able to speak, read and understand French
* Able to communicate by phone
* Written informed consent obtained from the patient
* Registration in a national health care system

Exclusion Criteria:

* Minor or protected adult
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of using oncological supportive cares after evaluation of supportive care needs reviewed by a professional of health, by a phone call | 4 to 6 weeks after baseline
  Assess the percentage of using oncological supportive cares after evaluation of supportive care needs reviewed by a professional. The use of supportive cares is evaluated with an hetero-questionnaire created for this study. The hetero-questionnaire consists in a phone call to evaluate the evolution of each item of the self-assessment questionnaire (which includes 6 evaluations : a nutritional evaluation (10 items), a social evaluation (8 items), a psychologic evaluation (6 items), a physiological evaluation (7 items), a pain evaluation (4 items) and a supportive care needs evaluation (6 items)).

SECONDARY OUTCOMES:
Evaluation of initial supportive care needs by the self-assessment questionnaire | baseline
  Assess the percentage of initial supportive care needs evaluated by the self-assessment questionnaire created for this study. It includes evaluations : a nutritional evaluation (10 items), a social evaluation (8 items), a psychologic evaluation (6 items), a physiological evaluation (7 items), a pain evaluation (4 items) and a supportive care needs evaluation (6 items).
Assess the correlation between supportive care needs and age | This analyse will be realized at the end of the study (9 weeks after baseline)
  Correlate the percentage of supportive care needs to age by a Pearson Chi squared test
Assess the correlation between supportive care needs and sexe | This analyse will be realized at the end of the study (9 weeks after baseline)
  Correlate the percentage of supportive care needs to sexe by a Pearson Chi squared test.
Assess the correlation between supportive care needs and type of cancer | This analyse will be realized at the end of the study (9 weeks after baseline)
  Correlate the percentage of supportive care needs to the type of cancer by a Pearson Chi squared test
Compare the percentage of using a supportive care professional judgement in regard to read and unread questionnaires by medical staff | This analyse will be realized at the end of the study (9 weeks after baseline)
  Assess the percentage of using a supportive care when the medical staff read the completed questionnaire. Assess the percentage of using a supportive care when the medical staff didn't read the completed questionnaire. Then compare these values by using a T- test of Student.
Compare the percentage of using a supportive care professional judgement in regard to the function of the medical staff member | This analyse will be realized at the end of the study (9 weeks after baseline)
  Assess the percentage of using a supportive care when the medical staff who read the completed questionnaire is a doctor, a nurse, or an auxiliary nurse . Then compare these values by using a T- test of Student
Assess the percentage of requirement to the physician during the study | 4 to 6 weeks after baseline (by a phone call, at the same time than the hetero-questionnaire)
  Assess the percentage of requirement to the physician during the study by asking each patient (by phone call)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique FRASIE, Md, Principal Investigator — Centre Paul Strauss
Locations (1):
- Centre Paul Strauss, Strasbourg, France